CLINICAL TRIAL: NCT07324369
Title: The Effect of Preoperative Education Based on ERAS Protocols on Postoperative Recovery in Patients Undergoing Colorectal Surgery: A Randomized Controlled Trial
Brief Title: Effect of Preoperative ERAS Education on Recovery After Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Deniz Şanlı, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0099
Record Dates: First submitted 2025-12-09; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: enhanced recovery after surgery; colorectal cancers; colorectal surgery; patient education; preoperative care
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study used a two-arm, parallel assignment randomized controlled design. Participants were individually randomized in a 1:1 ratio to either the intervention group, which received ERAS-based preoperative education, or the control group, which received standard preoperative care. Randomization was performed using a computer-generated sequence, and allocation was concealed with sealed opaque envelopes. The study was conducted as a single-blind trial in which the outcomes assessor (statistician) was blinded to group assignment.
Who Masked: Outcomes Assessor
Masking Description: Only the statistician performing the data analysis was masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS-Based Preoperative Education (Experimental): A structured preoperative education intervention based on ERAS recommendations for colorectal surgery. The session includes key components of preoperative, intraoperative, and postoperative care and is delivered once within 48 hours before surgery. A written educational booklet is provided to support patient understanding.
  Interventions: Behavioral: ERAS-Based Preoperative Education
- Standard Preoperative Education (Active Comparator): Routine preoperative education delivered by the ward nurse as part of the hospital's standard surgical preparation practices. No ERAS-based materials or additional educational content are included.
  Interventions: Behavioral: Standard Preoperative Education

INTERVENTIONS:
Behavioral: ERAS-Based Preoperative Education — A structured, individualized preoperative education session based on ERAS recommendations for colorectal surgery. The education includes information on preoperative, intraoperative, and postoperative practices. It is delivered by the researcher in a single 20-minute session within 48 hours before surgery (excluding the last 24 hours) and supported with a written educational booklet.
  Arms: ERAS-Based Preoperative Education
Behavioral: Standard Preoperative Education — Routine preoperative education provided by the ward nurse as part of the hospital's standard surgical preparation process. This education reflects usual care and does not include ERAS-based content or additional materials.
  Arms: Standard Preoperative Education

SUMMARY:
This randomized controlled trial describes the design and conduct of ERAS-based preoperative education in patients with colorectal cancer undergoing colorectal surgery. The study is conducted in the general surgery clinics of Izmir City Hospital. Eligible patients are randomly assigned to either an intervention group receiving structured preoperative ERAS-based education supported by an educational booklet or a control group receiving standard preoperative care routinely provided in the clinic.

Postoperative recovery outcomes are predefined in the study protocol. The primary outcome is postoperative recovery on the first postoperative day, measured using the Quality of Recovery-40 (QoR-40) questionnaire. Secondary outcomes include postoperative hospital length of stay, total length of hospital stay, reoperation during hospitalization, and 30-day readmission related to postoperative complications.

DETAILED DESCRIPTION:
Recovery following major colorectal surgery is a multidimensional process that includes physical, physiological, psychological, and functional components. Patients undergoing colorectal surgery may experience symptoms such as pain, discomfort, reduced mobility, and anxiety during the perioperative period. Enhanced Recovery After Surgery (ERAS) protocols provide a structured, evidence-based framework for perioperative care, within which patient education is included as part of the perioperative care process.

This randomized controlled trial describes the design and implementation of ERAS-based preoperative education for patients hospitalized with colorectal cancer and scheduled for colorectal surgery, with postoperative recovery outcomes predefined in the study protocol. The study is conducted in six general surgery clinics of Izmir City Hospital between January 2025 and November 2025. Patients who meet the inclusion criteria are randomly assigned to either an intervention group receiving structured preoperative education or a control group receiving standard preoperative instructions routinely provided in the clinic.

Randomization is performed using a computer-generated randomization list, and allocation is concealed using sealed opaque envelopes. The study is conducted as a single-blind trial in which patients are not informed of their group assignment. The researcher delivering the intervention and collecting the data is aware of group allocation, while statistical analysis is performed by an independent statistician without access to group assignment information.

Intervention Description:

The intervention consists of individualized preoperative education delivered in the patient's hospital room within 48 hours prior to surgery, but not within the final 24 hours before surgery. The educational content is based on ERAS recommendations for elective colorectal surgery and includes information related to perioperative care processes, such as nausea and vomiting prevention, preoperative fasting and carbohydrate intake, antibiotic prophylaxis, skin and bowel preparation, anesthesia and fluid management, temperature management, surgical approach, postoperative pain management, early nutrition and mobilization, catheter and drain management, blood glucose control, and recognition of potential postoperative complications.

The education session lasts approximately 20 minutes and is delivered using explanation, discussion, and question-and-answer techniques. Participants in the intervention group are provided with an educational booklet developed by the researcher, written in clear and accessible language, which serves as supplementary written material for review.

Control Group:

Participants in the control group receive standard preoperative education routinely provided in the clinic as part of the usual preoperative preparation process.

Outcome Measures:

The primary outcome is postoperative recovery on the first postoperative day, assessed using the Quality of Recovery-40 (QoR-40) questionnaire. Secondary outcomes include postoperative hospital length of stay, total length of hospital stay, reoperation due to postoperative complications, and 30-day readmission related to postoperative complications.

Data Collection:

Participants are visited by the researcher during the preoperative period (24-48 hours before surgery) and on the first postoperative day. Data are collected through face-to-face interviews using standardized data collection instruments, and relevant clinical information is obtained from medical records. Information regarding 30-day readmission is retrieved from electronic hospital databases following discharge.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Age 18 years or older
* Being literate
* Ability to understand and speak Turkish
* No diagnosed psychiatric disorder
* No cognitive impairment
* No visual or hearing impairment
* Being conscious, cooperative, and oriented
* Hospitalized with a diagnosis of colorectal cancer
* Scheduled to undergo colorectal surgery

Exclusion Criteria:

* Requirement for emergency surgery
* ASA score of IV or V
* Experiencing a serious complication during surgery
* Intraoperative creation of a stoma
* Admission to the intensive care unit after surgery
* Experiencing a serious postoperative complication
* Deterioration of general condition after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-40 (QoR-40) score on postoperative day 1 | Postoperative day 1 (24 hours after surgery)
  The QoR-40 questionnaire assesses postoperative recovery across five domains: emotional state, physical comfort, psychological support, physical independence, and pain. Higher scores indicate better quality of recovery. Total scores range from 40 to 200, with higher scores indicating better quality of recovery.

SECONDARY OUTCOMES:
Postoperative hospital length of stay | From the end of surgery through hospital discharge (up to 30 days)
  Number of days the patient remains hospitalized after surgery.
Total hospital length of stay | From the day of hospital admission through hospital discharge (up to 30 days)
  Total number of days hospitalized, including preoperative and postoperative days.
Reoperation due to postoperative complications | From the end of surgery through hospital discharge (up to 30 days)
  Occurrence of unplanned return to the operating room due to complications following the index surgery.
30-day hospital readmission due to complication | Within 30 days after discharge
  Readmission to the hospital caused by postoperative complications, as documented in electronic medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is a master's thesis project, and the informed consent form does not include permission for public data sharing. In addition, the dataset contains sensitive clinical information, and institutional policies do not allow disclosure of identifiable or de-identified patient data for external research use.